CLINICAL TRIAL: NCT02365740
Title: Postprandial Blood Glucose Control and Gastric Emptying in Patients With Type 1 Diabetes: Pathogenetic Factors, Clinical Relevance and Possible Therapeutic Options
Brief Title: Postprandial Blood Glucose Control and Gastric Emptying in Type 1 Diabetes: Pathogenetic Factors and Therapeutic Options
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Brunella Capaldo, MD, Federico II University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 248/13
Record Dates: First submitted 2015-02-04; First posted 2015-02-19 (Estimated); Last update posted 2015-02-19 (Estimated); Status verified 2014-11

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Type 1 Diabetes mellitus; Gastric Emptying; Insulin Infusion Pump
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Continuous Glucose Monitoring

ARMS (2):
- Cases (Experimental): gastric emptying test gut hormones determination Continuous Glucose Monitoring Insulin single bolus Insulin double-wave bolus
  Interventions: Other: gastric emptying test; Other: gut hormones determination; Other: Continuous Glucose Monitoring; Drug: Insulin single bolus; Drug: Insulin double-wave bolus
- Controls (Sham Comparator): gastric emptying test gut hormones determination
  Interventions: Other: gastric emptying test; Other: gut hormones determination

INTERVENTIONS:
Other: gastric emptying test — gastric emptying rate for solid will be determined using the 13C-OBT. Breath samples will be taken before the meal and then at 15-min intervals for a period of 240 min postprandially. The 13C content will be determined by on-line gas chromatographic purification-isotope ratio mass spectrometry (ABCA; Europe Scientific, Crewe, UK). The 13CO2 excretion curves will be analyzed and the half-emptying time (t½) and lag phase (tlag) calculated.
Other: gut hormones determination — blood sampling at 0, 15, 30, 60, 90, 120, 180 min for determination of plasma, glucagon and GI hormones (Ghrelin, GLP-1, GIP)
Other: Continuous Glucose Monitoring — 7 days Continuous Glucose Monitoring
  Arms: Cases
Drug: Insulin single bolus — pre-prandial insulin administered as single bolus calculated on the basis of carbohydrate counting and each patient's insulin/glycaemic load
  Arms: Cases
Drug: Insulin double-wave bolus — pre-prandial insulin fractioned into a double-wave bolus
  Arms: Cases

SUMMARY:
This study evaluates the prevalence of gastric emptying (GE) in type 1 diabetic patients (DM1) free of chronic complications in comparison with a group of healthy control subjects. The investigators will also assess the relationship between GE and glucose control (HbA1c, postprandial glucose variability), gut peptide hormones (GLP-1, GIP, and ghrelin), and gastrointestinal symptoms.

In addition, in patients with delayed GE the investigators will investigate the effect of "tailored" pre-prandial insulin bolus administered by means of insulin pump in reducing postprandial glucose variability, evaluated through continuous glucose monitoring system.

DETAILED DESCRIPTION:
Diabetic patients with a delayed GE will be studied in 2 separate occasions in euglycemic condition and under CGM. On both occasions, they will have to take a standard meal poor of lipids (rice 60 g; yellow squash 200 g; extra virgin olive oil 7 g; adult veal lean cuts 90 g; bananas 180 g; ordinary bread 75 g).

On the first occasion pre-prandial insulin will be administered as single bolus calculated on the basis of carbohydrate counting and each patient's insulin/glycaemic load.

On the second occasion the amount of pre-prandial insulin will be the same as the first one test but fractioned into a double-wave bolus. The "tailored" insulin bolus will be defined according to the individual pattern of GE, as follows:

* GE T1/2 121-180 min= 60% as bolus + 40% during following 2 h
* GE T1/2 >180 min= 40% as bolus + 60% during following 4 h Glycemic variability will be assessed by the means of Continuous Glucose Monitoring System and the following indexes of glucose variability will be calculated: number of hypoglycemic events, number of hyperglycemic events, standard deviation of glycemia, glycemia variation coefficient, mean range of daily glycemia, interquartile range, M value, mean amplitude of glycemic excursions (MAGE), low blood glucose index (LBGI), high blood glucose index (HBGI).

ELIGIBILITY:
Inclusion Criteria:

* DM1;
* Use of insulin pump;
* Disease duration ≥ 3 years.

Exclusion Criteria:

* Presence of chronic complications of DM (including cardiovascular autonomic neuropathy);
* BMI ≥ 30 kg/m2;
* Presence of chronic diseases other than DM1;
* Diseases that interfere with GE;
* Medications that interfere with blood glucose homeostasis (except insulin) and GE.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
gastric emptying measure | 4 hours

SECONDARY OUTCOMES:
gut hormones dosage | 3 hours
Continuous Glucose Monitoring | 7 days
postprandial glucose variability after single insulin bolus | 3 hours
postprandial glucose variability after double-wave insulin bolus | 3 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of "Medicina Clinica e Chirurgia" of Federico II University, Naples, Naples, Italy